CLINICAL TRIAL: NCT03015662
Title: Clinical Outcomes After Dry Needling on Cervical Muscles, Quality of Life, Fatigue, Quality of Sleep, Anxiety and Depression in Patients With Fibromyalgia Syndrome.
Brief Title: Clinical Outcomes After Dry Needling on Cervical Muscles, and Quality of Life, in Patients With Fibromyalgia Syndrome.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Almeria (Other)
Responsible Party: Principal Investigator, Adelaida María Castro-Sánchez, PhD, Full Professor, Universidad de Almeria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UAL-428
Record Dates: First submitted 2017-01-05; First posted 2017-01-10 (Estimated); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Fibromyalgia
Keywords: Quality of Life; Fatigue; Anxiety; Physical Therapy Modalities; Pain
MeSH Terms: conditions — Fibromyalgia; Fatigue; Anxiety Disorders; Pain | interventions — Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dry Needling Therapy (Experimental): Active or latent MTrPs (myofascial trigger points) will be remarked in black or red, respectively. Active or latent MTrPs will be needled in the same position employed by the blinded examiner for diagnosis. All dry needling procedures will be performed by the same investigator, and the technique used will be similar to the Hong method, using sterile Ener-Qi needles (EQ 1661) for the punction of TrPs (trigger points).
  Interventions: Other: Dry Needling Therapy
- Myofascial Release Therapy (Active Comparator): Patients will develope a myofascial therapy protocol, administered in the following order: deep fascia release in temporal region, suboccipital release, compression-decompression of temporomandibular joint, global release of cervicodorsal fascia, release of pectoral region, diaphragm release (transverse slide), and transverse diaphragmatic plane.
  Interventions: Other: Myofascial Release Therapy

INTERVENTIONS:
Other: Dry Needling Therapy — Dry needling procedures will be performed in the following pairs of muscles in the same intervention: occipital, splenius capitis, sternocleidomastoid (Clavicular branch TrPs 1, 2 and 3; sternal branch TrPs 1, 2, 3 and 4), scalene (anterior TrPs 1, and 2; medial TrP (Trigger Point) 1; posterior TrP 1), trapezius (upper TrPs 1, and 2; middle TrPs 5, 6 and 7; lower TrPs 3, and 4), supraspinatus (central point; myotendinous union; tendon insertion), infraspinatus (medial/superior; lateral/superior; lateral scapular side; medial scapular side), and multifidus (level C6).
  Arms: Dry Needling Therapy
Other: Myofascial Release Therapy — Patients will develope a myofascial therapy protocol, administered in the following order in the same intervention: deep fascia release in temporal region, suboccipital release, compression-decompression of temporomandibular joint, global release of cervicodorsal fascia, release of pectoral region, diaphragm release (transverse slide), and transverse diaphragmatic plane.
  Arms: Myofascial Release Therapy

SUMMARY:
Objectives: The purpose of the current randomized clinical trial is to compare the effectiveness of dry needling versus myofascial release therapy on myofascial trigger points (MTrPs) in cervical muscles, quality of life, fatigue, quality of sleep, anxiety and depression in patients with fibromyalgia syndrome (FMS).

DETAILED DESCRIPTION:
Design: A single-blind randomized controlled trial will be conducted on patients with FMS.

Methods: Sixty-four subjects with FMS will be randomly assigned to an experimental group receiving dry needling therapy, or to a control group for myofascial release therapy in the trigger points active or latent in the following pairs of muscles: occipital, splenius capitis, sternocleidomastoid, scalene, trapezius, supraspinatus, infraspinatus, and multifidus. Myofascial trigger points, quality of life, impact of fibromyalgia symptoms, quality of sleep, intensity of pain, anxiety levels, state of depression, impact of fatigue will be recorded at baseline and after four weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Fibromyalgia syndrome diagnosis.
* Aged from 18 to 60 years.
* No regular physical activity.
* Limitation of usual activities due to pain on at least 1 day in the previous 30 days.
* Agreement to attend evening therapy sessions

Exclusion Criteria:

* Receipt of any no pharmacologic therapies.
* Presence of cardiac, renal or hepatic insufficiency.
* Severe physical disability.
* Comorbid condition (eg, inflammatory disease).
* Infection fever.
* Hypotension.
* Skin alterations.
* Psychiatric illness.
* Previous history of surgery.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Active and Latent Myofascial Trigger Points (Number of trigger Points) | Change from baseline myofascial trigger points at four weeks
  Myofascial Trigger Points will be explored in the following pairs of muscles: occipital, splenius capitis, sternocleidomastoid, scalene, trapezius, supraspinatus, infraspinatus, and multifidus.

SECONDARY OUTCOMES:
Quality of Life (SF-36 quality of life questionnaire) | Change from baseline quality of life at four weeks
  The SF-36 quality of life questionnaire assesses 8 domains including physical functioning, physical role, bodily pain, general health, vitality, social functioning, role-emotional, and mental health.
Impact of Fibromyalgia Symptoms (Fibromyalgia Impact Questionnaire) | Change from baseline impact of fibromyalgia symptoms at four weeks
  The Spanish version of Fibromyalgia Impact Questionnaire (FIQ) will be used to assess the impact of FMS symptoms on physical and mental health of patients.
Quality of Sleep (Pittsburgh Quality of Sleep Questionnaire Index) | Change from baseline quality of life at four weeks
  The Pittsburgh Quality of Sleep Questionnaire Index (PSQI) will be used to study the quality of sleep. It comprises 24 items where the subjects respond to 19 of these items, and individual living in the same dwelling (or hospital room) responds to the remaining 5. Scores are obtained on each of 7 components of sleep quality: subjective quality, sleep latency, sleep duration, habitual sleep efficacy, sleep perturbations, use of hypnotic medication, and daily dysfunction.
Pain (Visual Analog Scale) | Change from baseline pain intensity at four weeks
  Pain will be assessed with the Visual Analog Scale (VAS), which assesses the pain intensity and degree of relief experienced by the patient (scored of 0 = no pain; 10 = unbearable pain).
Anxiety levels (State-Trait Anxiety Inventory ) | Change from baseline anxiety levels at four weeks
  Anxiety levels will be determined with the 40-item State-Trait Anxiety Inventory (STAI), which measures anxiety as a stable dimension of personality (trait or tendency to anxiety) and also includes a state subscale to detect anxiety behaviors.
State of depression (Beck Depression Inventory) | Change from state of depression at four weeks
  The state of depression will be determined with the Beck Depression Inventory (BDI), a self-applied 21-item questionnaire that assesses a wide spectrum of depressive symptoms. It focuses on the cognitive components of depression, which represent around 50% of the total questionnaire score.
Impact of fatigue (Fatigue Impact Scale ) | Change from impact of fatigue at four weeks
  The impact of fatigue will be determined with the Fatigue Impact Scale (FIS). It is a questionnaire-based inventory which requires patients to rate the perceived functional limitations about psychosocial, cognitive, and physical domains (with the maximum score of these sub-scales are 80, 40, and 40, respectively) due to fatigue over the previous month.

CONTACTS AND LOCATIONS:
Overall Officials: Adelaida María Castro-Sánchez, PhD, Principal Investigator — Universidad de Almeria
Locations (1):
- University of Almeria, Almería, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Castro-Sanchez AM, Mataran-Penarrocha GA, Arroyo-Morales M, Saavedra-Hernandez M, Fernandez-Sola C, Moreno-Lorenzo C. Effects of myofascial release techniques on pain, physical function, and postural stability in patients with fibromyalgia: a randomized controlled trial. Clin Rehabil. 2011 Sep;25(9):800-13. doi: 10.1177/0269215511399476. Epub 2011 Jun 14. PMID 21673013
- [Background] Montoya P, Pauli P, Batra A, Wiedemann G. Altered processing of pain-related information in patients with fibromyalgia. Eur J Pain. 2005 Jun;9(3):293-303. doi: 10.1016/j.ejpain.2004.07.012. PMID 15862479
- [Background] Vierck CJ Jr. Mechanisms underlying development of spatially distributed chronic pain (fibromyalgia). Pain. 2006 Oct;124(3):242-263. doi: 10.1016/j.pain.2006.06.001. Epub 2006 Jul 13. PMID 16842915
- [Background] Unverzagt C, Berglund K, Thomas JJ. DRY NEEDLING FOR MYOFASCIAL TRIGGER POINT PAIN: A CLINICAL COMMENTARY. Int J Sports Phys Ther. 2015 Jun;10(3):402-18. PMID 26075156
- [Background] Alonso-Blanco C, Fernandez-de-las-Penas C, Morales-Cabezas M, Zarco-Moreno P, Ge HY, Florez-Garcia M. Multiple active myofascial trigger points reproduce the overall spontaneous pain pattern in women with fibromyalgia and are related to widespread mechanical hypersensitivity. Clin J Pain. 2011 Jun;27(5):405-13. doi: 10.1097/AJP.0b013e318210110a. PMID 21368661
- [Background] Yeganeh Lari A, Okhovatian F, Naimi Ss, Baghban AA. The effect of the combination of dry needling and MET on latent trigger point upper trapezius in females. Man Ther. 2016 Feb;21:204-9. doi: 10.1016/j.math.2015.08.004. Epub 2015 Aug 14. PMID 26304789
- [Background] Hsieh YL, Kao MJ, Kuan TS, Chen SM, Chen JT, Hong CZ. Dry needling to a key myofascial trigger point may reduce the irritability of satellite MTrPs. Am J Phys Med Rehabil. 2007 May;86(5):397-403. doi: 10.1097/PHM.0b013e31804a554d. PMID 17449984
- [Background] Tough EA, White AR, Cummings TM, Richards SH, Campbell JL. Acupuncture and dry needling in the management of myofascial trigger point pain: a systematic review and meta-analysis of randomised controlled trials. Eur J Pain. 2009 Jan;13(1):3-10. doi: 10.1016/j.ejpain.2008.02.006. Epub 2008 Apr 18. PMID 18395479